CLINICAL TRIAL: NCT04028609
Title: Community Health Worker and Certified Peer Specialist Intervention to Improve Post-Hospital Outcomes
Brief Title: Community Health Worker Intervention to Improve Post-Hospital Outcomes
Acronym: CHW
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 prevented further enrollment
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency); Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Judith A. Cook, Professor of Psychiatry, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0715; 90RT5038a (Other Grant/Funding Number: National Institute Disability Independent Living Rehab)
Record Dates: First submitted 2019-07-11; First posted 2019-07-22 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Chronic Disease (Physical); Mental Disorder
Keywords: 30-day readmission; primary care; community health worker; health education
MeSH Terms: conditions — Chronic Disease; Mental Disorders; Health Education

STUDY DESIGN:
Intervention Model Description: The intervention includes 4 components: development of a personal health plan; review and support for medication adherence; connection with primary care provider within 30 days; and education about clinical indicators that call for immediate intervention.
Who Masked: Outcomes Assessor
Masking Description: Research interviewers were blinded to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects receive an intervention with 4 components: development of a personal health plan; review and support for medication adherence; connection with primary care provider within 30 days; and education about clinical indicators that call for immediate intervention.
  Interventions: Behavioral: Healthy at Home
- Services as Usual (Active Comparator): Subjects receive medical services as usual.
  Interventions: Other: Services as Usual

INTERVENTIONS:
Behavioral: Healthy at Home — In addition to receiving medical services as usual, subjects receive services from Community Healthy Workers during the transition from the hospital to their community residence.
  Arms: Intervention
Other: Services as Usual — Routine medical services
  Arms: Services as Usual

SUMMARY:
This study tests an intervention designed to avoid 30-day readmissions following a medical hospitalization by patients who have co-occurring mental illness. The Intervention is delivered by community health workers in the inpatient setting and 30 days following hospital discharge to the community.

DETAILED DESCRIPTION:
This study will test the efficacy of a brief intervention delivered to adults with co-occurring medical and mental health conditions by community health workers designed to avoid 30-day readmissions following medical hospitalization. Adult inpatients of a university hospital will be randomly assigned to the intervention plus services as usual versus services as usual alone, and assessed at baseline and 30 days following discharge. Chi square will be used to assess the primary outcome of admission within 30 days of discharge and changes in patient activation, mental health symptoms, medication adherence, and perceived competence for health maintenance. Also examined will be study condition differences in post-discharge inpatient service utilization and cost.

ELIGIBILITY:
Inclusion Criteria:

* receiving inpatient treatment for chronic medical condition
* evidence of a mental health diagnosis
* age 21- 60 years
* expected to return to community residence
* residing within a 30-mile radius of the hospital
* expected to remain in hospital for 2 or more days
* able to provide informed consent

Exclusion Criteria:

* terminally ill
* unable to communicate in English
* expected to be discharged to skilled facility or nursing home
* participating in another transitional care intervention
* hospitalized for behavioral health disorder

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Federal Center for Medicare and Medicaid Services' measure of unplanned readmissions that occur within 30 days of discharge from an initial admission | 30 days post discharge
  This is a dichotomous indicator variable that reports the occurrence of an inpatient admission to the hospital within 30 days of discharge from a previous hospitalization. Score ranges from 0 (no readmission) to 1 (readmission).
Federal Center for Medicare and Medicaid Services' measure of completion of a outpatient visit with primary care provider | during the 30 days period following discharge
  This is a dichotomous indicator variable that reports the completion of a patient's visit to an outpatient primary care provider

SECONDARY OUTCOMES:
Patient Activation Measure | study entry (pre-intervention), 30 days post discharge (post intervention)
  This scale measures the construct of a person's self-perceived ability to engage in health care. Items assess patients' self-perceived level of knowledge, skill, and confidence in their ability to manage their own health. Total score ranges from 13 to 52 with higher values indicating greater activation. Total score is calculated by summing items to create a raw score which is then divided by the number of items answered and multiplied by 13 and transformed to a Z score based on calibration tables.
Perceived Competence for Health Maintenance Questionnaire | study entry (pre-intervention), 30 days post discharge (post intervention)
  This scale measures the construct of self rated ability to manage one's health condition, engage in routine health care, and recover from a medical condition. Total score ranges from 1 to 7 with higher values indicating greater competence. Total score is calculated by averaging scores of the 4 items.
Short Form Health Survey | study entry (pre-intervention), 30 days post discharge (post intervention)
  This scale measures the construct of self-reported physical and emotional health by asking about functioning (e.g., climbing stairs, doing housework) and emotional well-being (e.g., feeling calm and peaceful, being downhearted or blue). Total score ranges from 12 to 44 with higher values indicating better health. Total score is the sum of all item responses.
Health Care Climate Questionnaire | study entry (pre-intervention), 30 days post discharge (post intervention)
  This scale measures the construct of a patients' perception of their medical care as as providing needed information, acknowledging their feelings, and supporting their autonomy. Total score ranges from 1 to 7 with higher values indicating greater autonomy. Total score is calculated by averaging the item scores.
Center for Disease Control and Prevention's National Health and Nutrition Examination Survey of Usual Source of Medical Care | study entry (pre-intervention), 30 days post discharge (post intervention)
  These items from a national household survey ask respondents about their access to and type of usual source of medical care. Both items are categorical self-report questions designed to yield descriptive information with no scoring.
Patient Satisfaction Questionnaire | study entry (pre-intervention), 30 days post discharge (post intervention)
  This a questionnaire that measures the construct of patients' satisfaction with their medical provider by asking them to rate their doctor's communication, time spent, and overall satisfaction. Total score ranges from 6 to 30 with higher values indicating greater satisfaction. Total score is calculated by adding the item scores.
Patient Health Questionnaire-2 | study entry (pre-intervention), 30 days post discharge (post intervention)
  This is a screening questionnaire for depression and anhedonia that measures the extent to which respondents report that they are sad, hopeless, and have little interest in doing things. Total score ranges from 0 to 6 with higher values indicating greater likelihood of depressive disorder. Total score is calculated by adding the 2 item scores.
Generalized Anxiety Disorder 2-item Questionnaire | study entry (pre-intervention), 30 days post discharge (post intervention)
  This is a screening questionnaire for generalized anxiety disorder that measures the extent to which respondents report that they are nervous, anxious, or continually worried. Total score ranges from 0 to 6 with higher values indicating greater likelihood of generalized anxiety disorder. Total score is calculated by adding the 2 item scores.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Cook, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Department of Psychiatry, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cook JA, Mueser KT. Community health workers: Potential allies for the field of psychiatric rehabilitation? Psychiatr Rehabil J. 2015 Sep;38(3):207-9. doi: 10.1037/prj0000164. PMID 26348316